CLINICAL TRIAL: NCT05616884
Title: A Prospective, Randomized Study Comparing Cemented and Cementless Fixed Bearing Unicondylar Medial Knee Replacement
Brief Title: Cemented vs. Cementless Unicompartmental Knee Arthroplasty
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Anderson Orthopaedic Research Institute (Other)
Responsible Party: Principal Investigator, Kevin B. Fricka, MD, Principal Investigator, Anderson Orthopaedic Research Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PRJ123
Record Dates: First submitted 2022-11-09; First posted 2022-11-15 (Actual); Last update posted 2023-07-24 (Actual); Status verified 2023-07

CONDITIONS: Partial Knee Replacement
Keywords: osteoarthritis; partial knee replacement; cementless
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Intervention Model Description: Prospective randomized trial, unblinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cementless (Experimental): Cementless fixation partial knee replacement
  Interventions: Procedure: Cementless fixation
- Cemented (Active Comparator): Cemented fixation partial knee replacement
  Interventions: Procedure: Cementless fixation

INTERVENTIONS:
Procedure: Cementless fixation — Three dimensional printed porous metal, a biomaterial with morphological and mechanical properties that resemble those of native trabecular bone, is now being used for fixation of the tibial component in unicondylar knee arthroplasty. This can reliably achieve osseointegration into the tibia and could lead to a lower risk of aseptic loosening which is the leading cause of revision in partial knee replacements.

SUMMARY:
The primary study objective is to evaluate a cementless partial knee system that has a modular 3-D printed porous metal tibial component and a cemented partial knee system. The hypothesis is that at minimum 2-year follow-up, fixed bearing medial partial knee replacements using cementless and cemented fixation will demonstrate no differences in clinical outcome.

DETAILED DESCRIPTION:
This is a prospective, randomized, unblinded clinical trial of 100 patients will be enrolled by invitation of the principal investigator. Inclusion criteria include patients 18-85 years old, patients receiving a medial fixed bearing partial knee replacement and patients deemed suitable for both cemented and cementless fixation after review of the preoperative radiographs. Minimum two-year outcome will be analyzed, and long-term follow-up will continue to 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Age18-85 years old
* medial fixed bearing partial knee replacement
* bone suitable for both cemented and cementless fixation after review of the preoperative radiographs.

Exclusion Criteria:

* Non-English speakers
* current smokers
* grossly porotic bone
* advanced other compartment arthritis at the time of surgery necessitating a total knee arthroplasty (TKA)
* previous high tibial osteotomy with prior hardware
* patients who are randomized but are deemed unsuitable to receive the assigned implant by the surgeon due to bone quality or bone cuts

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-07-08 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Knee Society Score | 2 years postoperative
  Clinical score for knee status and function. (0-100 scale, with 0 being the worst score and 100 being the best score.)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Hopper, Study Chair — Anderson Orthopaedic Research Institute
Locations (1):
- Anderson Orthopaedic Research Institute, Alexandria, Virginia, United States